CLINICAL TRIAL: NCT03205228
Title: Treatment Outcomes in Patients With Globus: A Randomized Control Trial of Psychoeducation, Anxiolytics and Proton Pump Inhibitors
Brief Title: Treatment in Patients With Globus: Psychoeducation, Anxiolytics or Proton Pump Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004/2560 (EC4)
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Globus
MeSH Terms: conditions — Globus Sensation | interventions — Omeprazole; Counseling; Palliative Care; flupentixol, melitracen drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flupentixol + Melitracen & placebo (Experimental): Deanxit® (Flupentixol + Melitracen) 5 mg/D*4 weeks will be given
  Interventions: Drug: Flupentixol +Melitracen
- Proton pump inhibitor & placebo (Active Comparator): Miracid® (Omeprazole) 20 mg/D*4 weeks will be given
  Interventions: Drug: Omeprazole
- Psychoeducation&placebo (Active Comparator): Psychoeducation by psychologists will be advised on Day 1 and Day 14 of the study time frame
  Interventions: Behavioral: psychoeducation

INTERVENTIONS:
Drug: Omeprazole — A capsule of Omeprazole 20 mg & 1 capsule of placebo will be given in individual subject, once daily for 4 weeks. Both drugs will be presented in the same appearance (white capsule).
  Other Names: Miracid®
  Arms: Proton pump inhibitor & placebo
Behavioral: psychoeducation — Psychoeducation will be given by psychologists at the Day 1 and Day 15 of the study period.One white capsule of placebo will be given once daily for 4 weeks of the study period.
  Other Names: advice for symptoms management
  Arms: Psychoeducation&placebo
Drug: Flupentixol +Melitracen — A capsule containing of a tablet of melitracen 10 mg + flupentixol 0.5 mg & a capsule of placebo will be given once daily, for 4 weeks. Both would be presented in the same appearance (white capsule)
  Other Names: Deanxit®
  Arms: Flupentixol + Melitracen & placebo

SUMMARY:
A randomized controlled trial study is conducted to compare treatment efficacy between psycho-education, anxiolytics drug and proton pump inhibitors in participants who met the criteria of globus.

DETAILED DESCRIPTION:
This is a randomized controlled trial in patients with globus. All participants will be allocated into 3 groups (16 subjects/group) : Proton pump inhibitors (miracid®) , anxiolytics drug (Deanxit®) and psycho-education. The study duration is 4 weeks long.

Data regarding clinical severity and quality of life of all participants will be collected at the beginning and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptoms based on the following criteria: Persistent or intermittent nonpainful sensation of a lump or foreign body in the throat with no structural lesion identified on physical examination, laryngoscopy, or endoscopy.

  1. Occurrence of the sensation between meals.
  2. Absence of dysphagia or odynophagia

Exclusion Criteria:

* Subjects with psychological disease
* Significant heart disease and/or arrhythmia
* Proton Pump inhibitors and/or Histamine 2 Receptor Antagonist use within 2 weeks before randomization
* Mono-amine Oxidase inhibitors or Selective Serotonin Reuptake Inhibitor or Tricyclic antidepressant use within 2 weeks before randomization
* History of drug allergy that use in research
* Pregnancy or breast feeding
* Decline to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-07-28 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 28 days
  Change in clinical scores assessed by Glasgow-Edinburgh throat Scale from baseline to the endo of the study

SECONDARY OUTCOMES:
Improvement in quality of life | 28 days
  Changes in the scores assessed by the 36-Item Short Form Health Survey questionnaire from baseline to the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Monthira Maneerattanaporn, MD., MS., Principal Investigator — Mahidol University
Locations (1):
- Division of gastroenterology, Department of Medicine, Siriraj hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No